CLINICAL TRIAL: NCT02220413
Title: Predictors and Moderators of Delayed Lactogenesis II and Duration of Breastfeeding
Brief Title: Predictors of Lactogenesis II
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 00018603
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-05

CONDITIONS: Breastfeeding
Keywords: Breastmilk; Lactogenesis; Obesity
MeSH Terms: conditions — Breast Feeding; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate what proportion of obese women will have a self-reported delay in lactogenesis II ("breastmilk coming in") compared to women with a normal weight. We hypothesize that obese women will have an absolute 20% increase in delayed lactogenesis II.

We will compare two group of women for delayed lactogenesis II, one group with obese women (BMI>30) and one group of women with a normal weight (BMI<30).

The secondary objective is to assess what other factors influence the self-reported delayed lactogenesis II.

DETAILED DESCRIPTION:
Lactogenesis I occurs during pregnancy (midpregnancy and beyond), when the mammary glands becomes sufficiently differentiated to secrete small quantities of specific milk components. Lactogenesis II is defined as the onset of plentiful milk secretion and typically occurs between 30-40 hours post delivery. It is typically described by women as a sense of fullness and leakage of milk which is subjectively reported between 50-73 hours post delivery. The incidence of delayed lactogenesis II ranges from 17-44%.

The risk of neonatal weight loss is up to 7 times greater for exclusively breastfed infants of women who experience delayed lactogenesis II as compared to women who experience typical onset lactogenesisII. In a qualitative study of 114 lactating women, increasing BMI was significantly associated with maternal perceptions of delayed onset of lactogenesis II.

The United States Breastfeeding Committee supports exclusive breastfeeding for the first 6 months of life because it "may exert a small but positive influence in reducing the risk of obesity in childhood and later in life…" Breastfeeding has also been associated with decreased risk of maternal morbidities such as type 2 diabetes, subclinical cardiovascular disease and less abdominal visceral adiposity. Given that prolonged breastfeeding improves the overall health of the mother infant dyad, it is critical to obtain a better understanding of those factors predictive of successful breastfeeding outcomes.

At University of South Florida our clinics serve an ethnically diverse population which would benefit from directed efforts at improving breastfeeding. Before we can undertake such a plan we need to assess the contemporary factors impacting lactogenesis.

We plan to prospectively enroll 186 pregnant women into a protocol to examine factors associated with delayed lactogenesis. Ninety-three women will have a BMI of 30 or higher at the time of delivery and the other 93 women will have a BMI ≤ 29 at the time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* intend to attempt breastfeeding
* Expecting a live-born infant
* Singleton pregnancy
* English or Spanish language fluency
* Delivered at fullterm gestation

Exclusion Criteria:

* Multiple gestation delivery
* Delivered pre-term (<36weeks and 6 days of gestation)
* Not admitted to Mother Baby Unit (MBU) (ie admitted to intensive or special care unit or to Labor & Delivery Unit for postpartum monitoring)
* Mother did not initiate breastfeeding within 12 hours.
* No telephone access
* History of breast reduction or enlargement surgery
* Planning to formula feed from birth (no intention to breastfeed or try breastfeeding).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We plan to prospectively enroll 186 pregnant women into a protocol to examine factors associated with delayed lactogenesis. Ninety-three women will have a BMI of 30 or higher at the time of delivery and the other 93 women will have a BMI ≤ 29 at the time of delivery.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Onset of lactogenesis II | 2-5 days post delivery
  Women will be asked about the perception of the onset of their breastmilk coming such as breast engorgement.

SECONDARY OUTCOMES:
Breastfeeding duration | Six weeks post delivery
  Women presenting for their 6 week postpartum exam will be asked to complete a short interview of 4 questions in regards to breastfeeding duration, "Measurement of intensity of breastfeeding behavior". Exclusivity of breastfeeding will be based on Labbok's suggested levels of breastfeeding behaviors.Women will be asked "How is your infant feeding? Why?" Responses will be categorized into exclusive, almost exclusive, partial high, partial low, token or no breastfeeding. Women not currently breastfeeding will be asked when the infant last received any breast milk and what the reason is for stop breastfeeding. If we miss the patient at their postpartum visit, we will complete the questionnaire by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Brumley, PhD, Principal Investigator — USF OB/GYN
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - USF South Tampa Center, Tampa, Florida
  - TGH Health Park Genesis Clinic, Tampa, Florida